CLINICAL TRIAL: NCT06972836
Title: Safety and Efficacy of Awake Uniportal Video Assisted Thoracoscopic Modified Pericardial Window in Recurrent Pericardial Effusion at Mid Term Result
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Elsayed Tawfek Ibrahim, assisstant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZU-IRB # 739-15-10-2024
Record Dates: First submitted 2025-04-24; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Awake Thoracoscope; Pericardial Effusion; Pericadiopleural Window
Keywords: pericardial effusion; pericardiopleural window
MeSH Terms: conditions — Pericardial Effusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake modified pericardial window (Experimental): H) shaped lines done by diathemy hoke above phrenic nerve then the upper and lower pericardial flabs reflelected outward in upper and lower directions respectively then 3 large clips applied on each angle of the reflected pericardial anlgles then heavy non absorbable suture is taken from the centre of the free reflected edge to adjacent upper and lower pericardium
  Interventions: Procedure: modified pericardial window
- General traditional pericardial window (Active Comparator): A portion of pericardium (2 cm diameter) was resected anterior to the phrenic nerve by diathermy hook
  Interventions: Procedure: traditional pericardial window

INTERVENTIONS:
Procedure: modified pericardial window — (H) shaped lines done by diathemy hoke above phrenic nerve then the upper and lower pericardial flabs reflelected outward in upper and lower directions respectively then 3 large clips applied on each angle of the reflected pericardial anlgles then heavy non absorbable suture is taken from the centre of the free reflected edge to adjacent upper and lower pericardium
  Arms: Awake modified pericardial window
Procedure: traditional pericardial window — A portion of pericardium (2 cm diameter) was resected anterior to the phrenic nerve by diathermy hook
  Arms: General traditional pericardial window

SUMMARY:
this study compare two surgical techniues at the same time two methods of anathesia with assisstance of thoracoscope for cases of repeated collection of fluid in pericardial sac and observation the result of the two techniques on the operated patients from 3 to 6 months

DETAILED DESCRIPTION:
this study compare two thoracoscopic techniues awake modified pericardial window and pericardial window under general anasethia for cases of repeated collection of fluid in pericardial sac and observation the result of the two techniques on the operated patients from 3 to 6 months

ELIGIBILITY:
Inclusion Criteria:

* patients who presented with recurrent massive pericardial effusion based on clinical, radiological evidence by Echo and C.T. chest

Exclusion Criteria:

* hemodynamically unstable patients

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
recurrence of pericardial effusion | follow up each month at out patient clinic for 6 months from the date of surgery
  clinical (Beck's triad:Hypotension with a narrowed pulse pressure,jugular venous distension,distant heart sounds )and Echo findings suggestive of recurrence of pericardial effusion
Awake anasethia | from the start till the end of the procedure about 45 min
  the patient is sedated -cooperative- hemodynamically stable by transthoracic spinal anasthsia at Cervical 5

CONTACTS AND LOCATIONS:
Overall Officials: Amr Tawfek, as prof, Principal Investigator — cardiothoracic surgery department-faculty of medecine-zagazig univeristy-Egypt
Locations (2):
- Egypt (2):
  - Amr El Sayed Tawfek, Zagazig, Sharqia Province
  - cardiothorathic surgery department -faculty of medecine-zagazig univeristy- Egypt, Zagazig, Sharqia Province

IPD SHARING:
Plan to Share IPD: No